CLINICAL TRIAL: NCT01076868
Title: Determining the Incidence of New Plasmodium Vivax Infections After Radical Treatment Following Vivax Malaria Along the Thai Burma Border
Brief Title: Incidence of Vivax Along the Thai Burma Border
Acronym: VHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SMRU0909
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2018-10

CONDITIONS: Vivax Malaria
Keywords: vivax; malaria; relapse
MeSH Terms: conditions — Malaria, Vivax; Malaria; Recurrence | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primaquine (Experimental): Primaquine 14 days
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — Primaquine x 14 days
  Other Names: primaquine 0.5 mg/kg/day

SUMMARY:
This is a continuous cohort study consisting of 200 participants (one third 6 months old to 5 years, one third 6 to 15 years old, one third ≥ 15 years old) i.e. a new patient will be recruited (from the same age group) for any patient who develops a Pv infection so that the cohort will always have 200 patients for 3 years. Each patient will be actively followed-up every 8 weeks until Plasmodium vivax infection occurs but the duration of follow up and the number of follow up visits for each patient will vary depending on when or if a vivax infection occurs and when the patient is recruited. Therefore, the minimum follow up period for each patient will be 6 months or time to vivax infection and the maximum will be 3 years if a patient does not get vivax infection and is recruited at the beginning of the study.

DETAILED DESCRIPTION:
This study will evaluate the most likely approach to malaria elimination; the administration of a radical curative dose of primaquine to the entire potentially infected population. In this study we will focus on patients who have had vivax malaria in the past year and so are very likely to harbour liver hypnozoites. Radical treatment is not given on the Thai-Burmese border because risks are considered to outweigh benefits, but it is recommended in Thailand. We believe that this policy could be changed if there was sufficient information.

Patients who have received chloroquine only treatment could be considered as incompletely treated. We plan to conduct a carefully documented evaluation of radical treatment in such patients. Through this we aim to determine the incidence of vivax malaria in patients living in a vivax endemic area following radical treatment. This will provide information on the safety and tolerability of primaquine, used in the context most likely during an elimination programme, and also will provide information on the incidence of vivax malaria. Adults and children > 6 months old with a documented P.vivax infection in the last 12 months will be recruited. In conjunction with a parallel study evaluating epidemiology in treated vivax malaria, we will be able to characterize the relapse history of P vivax. This will provide the foundation for further studies evaluating the efficacy of primaquine regimens.

Conclusions: The incidence of new Pv infection after radical cure with primaquine is estimated to be 0.2 infections/person year and declined during the course of the study. Further results have not been analysed yet.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic adults and children ≥ 6 months
* Documented P.vivax infection in the last 12 months who have not received radical treatment with primaquine
* Weight≥ 7 kg for children
* Participant (or parent/guardian if <18 years old) is willing and able to give written informed consent
* Ability (in the investigators opinion) and willingness of patient or parent/guardian to comply with all study requirements

Exclusion Criteria:

* History of allergy to primaquine
* Medical conditions such as known chronic diseases (TB, HIV, cardio vascular diseases), allergies, mental illnesses and similar conditions that could make the interpretation of symptoms or the follow up difficult.
* Other conditions such as drug addiction, known poor compliance with treatment or follow up.
* Inability to tolerate oral medication
* Pregnancy
* G6PD deficiency
* Blood transfusion in the last 3 months
* Microscopic evidence of Plasmodium vivax, P.falciparum, P. malariae or ovale
* Fever ≥37.5C

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2010-02; Primary Completion 2014-09-02 (Actual); Study Completion 2014-09-02 (Actual)

PRIMARY OUTCOMES:
Incidence | Up to 3 years
  Incidence of primary infections with vivax malaria

SECONDARY OUTCOMES:
Adverse events | Up to 3 years
  Adverse event profile of primaquine

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, MD, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand